CLINICAL TRIAL: NCT01201603
Title: The Effects of Orange Juice on Insulin Sensitivity and Plasma Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Florida Department of Citrus (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RIS 100058
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Insulin Resistance; Obesity
Keywords: Women; Orange Juice; Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orange Juice (Experimental): Orange Juice reconstituted from frozen concerntrate
  Interventions: Dietary Supplement: orange juice
- Orange drink (Placebo Comparator): Sugars matched orange drink
  Interventions: Dietary Supplement: orange juice

INTERVENTIONS:
Dietary Supplement: orange juice — 250ml of orange juice or a sugars matched orange drink

SUMMARY:
The aim of this study is primarily to investigate the ability of antioxidants found in orange juice (OJ) to increase the body's sensitivity to the hormone insulin. Overweight or mildly obese women, who are otherwise healthy, will be recruited. The time commitment for subjects is ~14wks. Subjects will attend the laboratory on 5 occasions after fasting from midnight. The 1st is a medical screening. Laboratory visits 2 & 5 will take ~5hrs and will be separated by 3 months, during which time subjects will consume 250ml of an orange drink (either OJ or an orange flavoured control drink) once a day. During visits 2 & 5, subjects will have a scan to assess their %body fat using a low-dose x-ray machine, and have their insulin sensitivity measured using a technique called a 'Glucose Clamp'. During the 3hr glucose clamp, subjects receive an infusion of the hormone insulin and a glucose solution directly into their blood stream, with insulin sensitivity determined from the amount of glucose required to maintain blood glucose at normal levels. In addition, a small sample of fat tissue (about the size of a haricot bean) will be taken from underneath the skin of the belly. Subjects will record their food intake for 3-days in weeks 3, 7 and 11 of consuming the drink, and come to the lab for visits 3&4 during weeks 4&8. Laboratory visits 3&4 repeat measurements taken in the 1st (screening) visit.

DETAILED DESCRIPTION:
Background:

Overweight and mild obesity are associated with insulin resistance and mild elevations in lipid risk factors which are not usually sufficiently abnormal to merit treatment. Such people are encouraged to lose weight to reduce their risk of progressing to type 2 diabetes and coronary heart disease, but there is clearly a potential role for dietary modifications to maximize any potential benefit of this weight loss. Flavonoids are known to have vascular effects which might enhance substrate delivery to metabolically active tissues, and thus improve insulin sensitivity. There are many different dietary sources of flavonoids, with fruits such as apples, berries and citrus being rich sources. However, some researchers have expressed concern that a high dietary intake of 100% juice may contribute to the development of insulin resistance, obesity and the Metabolic Syndrome (Bazzano, Li et al. 2008), although this is not universally accepted (Fujioka, Greenway et al. 2006; O'Neil and Nicklas 2008). To date, there have been no studies investigating the effects of citrus fruits on indices of cardio-metabolic health in people who are presently healthy but are at risk of developing some features of the Metabolic Syndrome.

Aims:

To investigate the effects of orange juice (OJ) intake on insulin sensitivity, appetite hormones, blood pressure and plasma lipids. In addition we aim to investigate any gene expression changes associated with OJ consumption, in particular in adipose tissue.

Experimental protocol and methods:

Overweight or obese women (BMI 27-35), who are otherwise healthy, will be recruited onto the study. They will attend the 'David Greenfield Human Physiology' laboratories on 5 convenient mornings, following an overnight fast. The 1st visit is a medical screening and will involve signing a consent form, completing medical screening, food frequency and activity questionnaires, having height, weight, and hip/waist circumference measurements taken and a sample of blood taken for CBC, urea, electrolytes, LFT, TFT, glucose and insulin analysis. Subjects will then be asked to complete a 3-day diet diary for macronutrient assessment and to consume a diet providing 50% of energy as carbohydrate for 3 days prior to the 2nd laboratory visit. This 2nd visit will involve having a DEXA body composition scan, an adipose tissue biopsy and a 3-hr hyperinsulinemic, euglycemic glucose clamp. Starting on the following morning, subjects will then consume an orange drink (either OJ or a carbohydrate matched orange flavoured drink) once a day for 12 wks. A 3-day diet diary for macronutrient assessment will be recorded during wks 3,7and 11 of taking the drink, and measurements made at screening will be repeated on visits 3 and 4 which will take place in weeks 4 and 8. A standardized diet will be consumed for 3 days prior to the final laboratory visit, as before. This 5th visit will be identical to visit 2.

ELIGIBILITY:
Inclusion Criteria:

* pre-menopausal or post-menopausal and taking HRT
* BMI 27-35kg/m2
* HOMA-IR value > 1.5
* healthy

Exclusion Criteria:

* pregnant or breast feeding,
* any metabolic or endocrine abnormalities,
* clinically significant abnormalities on screening,
* fasting glucose > 6.0mmol/l,
* taking medication other than the contraceptive pill or HRT
* herbal supplement use,
* food allergies/intolerances related to the investigational product (citrus juices, fructose)
* daily consumption of >100ml citrus juices

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity ('M' value) | after 3 months' intervention
  Insulin sensitivity (mg glucose disposal from the blood/kg body weight/min)calculated from glucose disposal during a hyperinsulinemic, euglycemic glucose clamp

SECONDARY OUTCOMES:
Glucose Oxidation rate | after 3 months' intervention period
  Measured by ventilated hood indirect calorimetry
High Density Cholesterol | after 3 months' intervention
  Serum HDL concentration
Low density cholesterol | after 3 months' intervention
  Serum LDL concentration
Gene expression in adipose tissue | after 3 months' intervention
  Expression of genes related to insulin sensitivity in adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bazzano LA, Li TY, Joshipura KJ, Hu FB. Intake of fruit, vegetables, and fruit juices and risk of diabetes in women. Diabetes Care. 2008 Jul;31(7):1311-7. doi: 10.2337/dc08-0080. Epub 2008 Apr 4. PMID 18390796
- [Background] Fujioka K, Greenway F, Sheard J, Ying Y. The effects of grapefruit on weight and insulin resistance: relationship to the metabolic syndrome. J Med Food. 2006 Spring;9(1):49-54. doi: 10.1089/jmf.2006.9.49. PMID 16579728
- [Background] O'Neil CE, Nicklas TA. A review of the relationship between 100% fruit juice consumption and weight in children and adolescents. American Journal of Lifestyle Medicine 2(4): 315-354, 2008.